CLINICAL TRIAL: NCT00006190
Title: The Study of Mechanisms of Lipodystrophy in HIV-Infected Patients
Brief Title: A Study to Determine How and Why HIV-Infected Subjects on Anti-viral Treatment Develop Lipodystrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: Double | Purpose: Diagnostic
Other Study IDs: lipod (completed); R01DK056583-01 (NIH)
Record Dates: First submitted 2000-08-25; First posted 2000-08-28 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: Lipoproteins; Insulin resistance; Adipose tissue
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Insulin Resistance | interventions — Nelfinavir; Stavudine; Lamivudine; efavirenz

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Stavudine
Drug: Lamivudine
Drug: Efavirenz

SUMMARY:
HIV infection is a major global health problem. Survival and quality of life for HIV subjects has tremendously improved with the advent of a class of antivirals called protease inhibitors and the utilization of highly active combination therapy. However, such therapy has been associated with a syndrome called lipodystrophy. This lipodystrophy syndrome causes body shape changes; typically thinning and loss of fat from the arms, legs and face, with increased fat appearing in the abdomen and neck. There are also metabolic changes which occur, and subjects can develop increased triglycerides, increased cholesterol and an increased risk for diabetes as indicated by increasing insulin resistance. This study will take HIV positive subjects who have not yet started antiviral medications (treatment naive)and randomly assign them to one of two treatment arms. These treatment arms will be: Sustiva/Zerit/Epivir vs. Viracept/Zerit/Epivir The subjects will be treated and followed for two years and have extensive metabolic testing, skinfold thickness measurements, MRI scans and other measures to determine if and how they are experiencing changes in metabolism or body shape and to discover the mechanism of why this occurs. Understanding the mechanism should allow researchers to design interventions for subjects who have lipodystrophy and strategies to prevent lipodystrophy from occurring to subjects treated with antivirals in the future.

ELIGIBILITY:
Inclusion Criteria:

* CD4 count > 200 cells/mm
* HIV RNA (viral load) <= 100,000 copies/ml
* No previous antiviral therapy

Exclusion Criteria:

* AIDS or opportunistic infections
* Active intravenous drug users
* Use of: corticosteroids, androgens, lipid-lowering drugs, anti-fungal medications, oxandrolone, megace, dehydroepiandrosterone.
* Subjects with diabetes mellitus
* Subjects who consume > 2 alcoholic drinks per day
* Pregnant women, premenopausal women unless adequate birth control is in use.
* Acute or chronic liver diseases, liver enzymes elevations > 2.5 times the upper limit of normal.
* Anemia, an Hct < 35% for men, or < 32% for women.
* Abnormal thyroid function tests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Abhimanyu Garg, Principal Investigator — University of Texas Southwestern Medical Center; Dr. Dolores Peterson — University of Texas Southwestern Medical Center; Dr. Ruth Berggren — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hengel RL, Watts NB, Lennox JL. Benign symmetric lipomatosis associated with protease inhibitors. Lancet. 1997 Nov 29;350(9091):1596. doi: 10.1016/s0140-6736(05)64011-1. No abstract available. PMID 9393341
- [Background] Carr A, Samaras K, Burton S, Law M, Freund J, Chisholm DJ, Cooper DA. A syndrome of peripheral lipodystrophy, hyperlipidaemia and insulin resistance in patients receiving HIV protease inhibitors. AIDS. 1998 May 7;12(7):F51-8. doi: 10.1097/00002030-199807000-00003. PMID 9619798
- [Background] Viraben R, Aquilina C. Indinavir-associated lipodystrophy. AIDS. 1998 Apr 16;12(6):F37-9. doi: 10.1097/00002030-199806000-00001. PMID 9583592
- [Background] Shaw AJ, McLean KA, Evans BA. Disorders of fat distribution in HIV infection. Int J STD AIDS. 1998 Oct;9(10):595-9. doi: 10.1258/0956462981921189. PMID 9819110
- [Background] Kotler DP, Rosenbaum K, Wang J, Pierson RN. Studies of body composition and fat distribution in HIV-infected and control subjects. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Mar 1;20(3):228-37. doi: 10.1097/00042560-199903010-00003. PMID 10077170
- [Background] Lo JC, Mulligan K, Tai VW, Algren H, Schambelan M. "Buffalo hump" in men with HIV-1 infection. Lancet. 1998 Mar 21;351(9106):867-70. doi: 10.1016/S0140-6736(97)11443-X. PMID 9525364